CLINICAL TRIAL: NCT06112574
Title: Enhancing Recovery in Stroke Through Combined Cognitive-motor Training - a Randomized Controlled Trial
Brief Title: Cognitive-motor Training Post-stroke - a Pilot Randomized Controlled Trial
Acronym: Cogmos
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Danderyd Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COGMOS-pilotRCT
Record Dates: First submitted 2023-09-11; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Stroke Sequelae; Motor Skills Disorders
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-task (Active Comparator): Visuomotor training
  Interventions: Behavioral: Visuomotor force control training
- Dual-task (Experimental): Visuomotor + cognitive components training
  Interventions: Behavioral: Visuomotor force control training

INTERVENTIONS:
Behavioral: Visuomotor force control training — Single-task training involves visuomotor finger force tracking and dual-task has an additional cognitive components including visual distraction and working memory.

SUMMARY:
Stroke is a leading and growing cause of long-term adult disability. Up to 80% of stroke patients have impaired manual dexterity reducing their independence, return to work and quality of life. Cognitive impairment is also common after stroke and growing evidence suggests a cognitive-motor interdependence with relevance for motor recovery. Previous studies show increased cognitive-motor interference (measured in dual-task) in stroke patients and that combining motor and cognitive task training (in a dual-task) may improve motor function above that achieved by single-task training. This project addresses post-stroke dexterity impairment and its relation to dual-task interference, i.e., the decrease in motor performance when performing a concurrent cognitive task. The overall goal is to provide a proof-of-concept for a dual-task interference training protocol post-stroke. We aim to establish therapeutic efficacy of dual-task vs single-task dexterity training in chronic stroke patients.Single-task training involves visuomotor finger force tracking and dual-task has an additional cognitive components including visual distraction and working memory. Training will be done 4 days/week over four weeks (total 16 sessions). Each session will include 20 mins of conventional therapy (stretching, functional exercises) followed by 40 mins motor task training (either single or dual task). This pilot randomized clinical trial will include 40 stroke patients (> 6 months after stroke). Repeated clinical and fine-grained motor measurements will be obtained pre and post intervention and at 3 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* adults with clinical diagnosis of stroke and history of upper limb hemiparesis. Arm and hand paresis is defined as weakness according to Manual Muscle Testing (score less than 4/5 in one upper limb muscles)
* reported difficulty in opening/closing of hand or difficulty in using the hand in daily activities

Exclusion Criteria:

* inability to grasp and displace an object (minimum score of 1 on Box and Block Test, BBT)
* impaired cognition (MOCA score <23)
* cerebellar stroke
* aphasia disturbing communication and understanding of training task
* neglect interfering with ability to see task on screen

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment change (FMA change) | At baseline and at 3 to assess change.
  Assesses sensory and movement related functions in the upper extremity (0 points max impairment summed up to 66 points max no detected impairment)

SECONDARY OUTCOMES:
Box and Block change (BBT change) | At baseline and at 3 to assess change.
  Assesses gross dexterity by timing how many blocks can be grasped and displaced in one minute (measured as blocks/min)
Logical reasoning change (WAIS IV matrices change) | At baseline and at 3 to assess change.
  Assesses intelligence through four composite socres: verbal comprehension, perceptual reasoning, working memory and processing speed (scored from 45 to 155).
Attention change (D-KEFS trail making test 1-5) | [At baseline and at 3 to assess change.
  Trail making test assesses attention capacites in five conditions: visual scanning, number sequencing, letter sequencing, number-letter sequencing, and motor speed (the speed of each condition is noted in seconds, max 150seconds).
Executive function change (D-KEFS FAS, D-KEFS tower) | At baseline and at 3 to assess change.
  Assesses executive function capacities such as spatial planning, rule learning, inhibition of impulsive responding, inhibition of perseverative responding, and establishing and maintaining instructional set. Scoring: raw scores are converted to scaled scores through established age and gender normative data, Mean=10, standard deviation=3).

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Danderyd Hospital, Division of Rehabilitation Medicine, Dept. of Clinical Sciences, Karolinska Institutet, Stockholm, Danderyd
  - Department of Rehabilitation Medicine, Danderyd Hospital, Danderyd, Stockholm County

IPD SHARING:
Plan to Share IPD: No